CLINICAL TRIAL: NCT00172380
Title: Phase II Study Evaluating Docetaxel and CDDP as Neoadjuvant Chemotherapy Prior to Surgery, Followed by Adjuvant Docetaxel Plus CDDP in Chemonaive Patients With NSCLC Stage III
Brief Title: Phase II Study of Docetaxel Plus CDDP for NSCLC Stage III
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 930911
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: NSCLC
MeSH Terms: interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- docetaxel and cisplatin (Experimental): docetaxel 36mg/m2 and cisplatin 75mg/m2
  Interventions: Drug: Docetaxel Plus CDDP

INTERVENTIONS:
Drug: Docetaxel Plus CDDP — docetaxel 36mg/m2 and cisplatin 75mg/m2

SUMMARY:
To assess the overall response rate to docetaxel plus CDDP as neoadjuvant chemotherapy prior to surgery, followed by adjuvant docetaxel plus CDDP in chemonaive patients NSCLC Stage IIIa and IIIb.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed NSCLC, respectable NSCLC stage IIIa T1-2 N2 or or unresectable stage IIIb 2.KPS>70% 3.Hb>10g/dl,ANC>2.0x109/L,Plt.>100x109/L4.T-bil.<1xULN,creatinine<1xULN,creatinine clearance >60 ml/min,GPT/GOT<2.5xULN,ALP<5xULN

Exclusion Criteria:

* 1.Brain meta.2..Prior surgery,R/T, C/t or immunotherapy for NSCLC

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2005-02; Primary Completion 2010-01 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
overall response rate | every cycle during 2nd-6th cycles

SECONDARY OUTCOMES:
resectability | resectability after treatment
progression free survival | progression free survival after 1 year
overall survival | overall survival at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Chong-Jen Yu, M.D,Ph.D., Principal Investigator — Department of Internal Medicine, National Taiwan University hospital
Locations (1):
- Department of Internal Medicine, National Taiwan University Hospital, Taipei, Taiwan